CLINICAL TRIAL: NCT06494215
Title: Comparison of Different Methods to Calculate Pendelluft by Electrical Impedance Tomography in Patients Undergoing Invasive Mechanical Ventilation Under Pressure Support Mode
Brief Title: Comparison of Different Methods to Calculate Pendelluft by Electrical Impedance Tomography in Mechanically Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 79317924.0.0000.0068
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Asynchrony, Patient-Ventilator; ARDS; Respiratory Insufficiency; Respiratory Effort-Related Arousal | Patient | Respiratory Measures and Ventilator Management
Keywords: Pendelluft; Ventilator-patient asynchrony; Patient self-induced lung injury; ARDS; Respiratory failure; Electrical Impedance Tomography
MeSH Terms: conditions — Patient-Ventilator Asynchrony; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: All the participants shall be exposed to the same situations (variation of pressure support and inspiratory/expiratory pauses)
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pressure Support Variation (Other): Patients shall be submitted to pressure support variation in a randomly assigned manner. First 30 minutes after plethysmogram stabilization shall be recorded at clinical pressure support. Next, a blood gas sample shall be collected by a nurse or a physician, and three inspiratory pauses of at least 2 seconds shall be performed in between eight respiratory cycles. Next three expiratory pauses shall be performed in between eight respiratory cycles. All data shall be recorded and analysed offline. Subsequently the same sequence of events shall be performed at a 50% higher pressure support and at a 50% lower pressure support. The sequence in which this will happen shall be randomly assigned (first lower PS vs higher PS or first higher PS vs lower PS).
  Interventions: Other: Pressure Support Variation and Calculation of Respiratory Mechanics

INTERVENTIONS:
Other: Pressure Support Variation and Calculation of Respiratory Mechanics — Patients will be submitted to different levels of pressure support (PS) in a randomly assigned order. First 30 minutes shall be recorded at the clinical PS. Next, blood gas samples shall be collected. Subsequently, three inspiratory pauses of at least 2 seconds shall be performed with an interval of at least 8 respiratory cycles between them. The same shall be performed with three expiratory pauses. Next, the PS shall be varied to 50% less or 50% more than clinical PS (based on randomization) and the same procedures shall be performed after 30 minutes of data recording (blood gas sample collection, inspiratory and expiratory pauses). All data shall be analyzed offline using a software that will be able to compare three different methods to calculate Pendelluft magnitude based on the literature. After completion of the protocol, ventilatory parameters shall be returned to the original settings. If the patient becomes tachypneic during lower PS, the protocol shall be interrupted.

SUMMARY:
The Pendelluft phenomenon is an important cause of lung damage in spontaneously breathing mechanically ventilated patients since it considerably increases the stress on the lung parenchyma in the dependent areas. It can result in a local driving pressure up to three times higher than the global driving pressure. The measurement of Pendelluft is still uncertain in the literature, and although various methods have been proposed, not all have the same meaning in terms of pulmonary overstress and overstrain. This study proposes a comparative analysis of different ways to calculate and estimate the stress imposed on the lung parenchyma by Pendelluft in terms of regional volume and local driving pressure through electrical impedance tomography.

DETAILED DESCRIPTION:
Respiratory mechanics and regional ventilation will be monitored by electrical impedance tomography (Enlight 1800 and 2100, Timpel). Esophageal and gastric pressures will be obtained by placing an esophageal/gastric balloon cathether (Nutrivent ®), validation concerning position will be done through modified Baydur maneuver (delta esophageal/delta airway pressure = 0.8-1.2). The hardware Pneumodrive will be used to inflate the balloon and store the airway, gastric and esophageal pressures.

Initially the patients will be monitored with EIT for aproximately 30 minutes after pletismography stabilization. Then, an arterial blood-gas sample shall be collected for analysis. Next, three expiratory and three inspiratory pauses of at least two seconds will be realized with intervals of eight respiratory cycles between them, allowing plateau pressure to be recorded and global and regional driving pressure to be estimated. All this data will be stored for later analysis. The same procedures and measurements shall be made sequentially with a 50% higher pressure support and with a 50% lower pressure support.

ELIGIBILITY:
Inclusion Criteria:

* Patients under invasive mechanical ventilation intubated due to respiratory failure in pressure support mode (weaning phase)

Exclusion Criteria:

* Age less than 18 years; sedation or neuromuscular blockade; absence of respiratory effort; contraindications to esophageal balloon cathether positioning or electrical impedance tomography belt positioning; presence of pneumothorax or active air leaks; hemodynamic instability; absence of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-06-11 (Estimated)

PRIMARY OUTCOMES:
1. Magnitude of Pendelluft | During 30 minutes after plethysmogram stabilization at clinical PS, during 30 minutes at 50% lower PS, and during 30 minutes at 50% higher PS
  Three differents methods of estimating magnitude of Pendelluft shall be compared using a software based on electrical impedance tomography monitoring (Enlight 2100, Timpel Medical®, Brazil)
2. Magnitude of Pendelluft during inspiratory pause | During 30 minutes after plethysmogram stabilization at clinical PS, during 30 minutes at 50% lower PS, and during 30 minutes at 50% higher PS
  One of the methods of Pendelluft measurement shall be performed during an inspiratory pause for comparison with a normal cycle (without pause).
3. Magnitude of respiratory effort | During 30 minutes after plethysmogram stabilization at clinical PS, during 30 minutes at 50% lower PS, and during 30 minutes at 50% higher PS
  Respiratory effort shall be estimated through expiratory pauses and though recording of esophageal pressure at different pressure support levels. These data shall be compared to Pendelluft magnitude according to the different methods of calculation

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo BP Amato, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Putensen C, Zech S, Wrigge H, Zinserling J, Stuber F, Von Spiegel T, Mutz N. Long-term effects of spontaneous breathing during ventilatory support in patients with acute lung injury. Am J Respir Crit Care Med. 2001 Jul 1;164(1):43-9. doi: 10.1164/ajrccm.164.1.2001078. PMID 11435237
- [Background] Sassoon CS, Zhu E, Caiozzo VJ. Assist-control mechanical ventilation attenuates ventilator-induced diaphragmatic dysfunction. Am J Respir Crit Care Med. 2004 Sep 15;170(6):626-32. doi: 10.1164/rccm.200401-042OC. Epub 2004 Jun 16. PMID 15201132
- [Background] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. Spontaneous breathing during lung-protective ventilation in an experimental acute lung injury model: high transpulmonary pressure associated with strong spontaneous breathing effort may worsen lung injury. Crit Care Med. 2012 May;40(5):1578-85. doi: 10.1097/CCM.0b013e3182451c40. PMID 22430241
- [Background] Yoshida T, Fujino Y, Amato MB, Kavanagh BP. Fifty Years of Research in ARDS. Spontaneous Breathing during Mechanical Ventilation. Risks, Mechanisms, and Management. Am J Respir Crit Care Med. 2017 Apr 15;195(8):985-992. doi: 10.1164/rccm.201604-0748CP. PMID 27786562
- [Background] Yoshida T, Torsani V, Gomes S, De Santis RR, Beraldo MA, Costa EL, Tucci MR, Zin WA, Kavanagh BP, Amato MB. Spontaneous effort causes occult pendelluft during mechanical ventilation. Am J Respir Crit Care Med. 2013 Dec 15;188(12):1420-7. doi: 10.1164/rccm.201303-0539OC. PMID 24199628
- [Background] Arellano DH, Brito R, Morais CCA, Ruiz-Rudolph P, Gajardo AIJ, Guinez DV, Lazo MT, Ramirez I, Rojas VA, Cerda MA, Medel JN, Illanes V, Estuardo NR, Bruhn AR, Brochard LJ, Amato MBP, Cornejo RA. Pendelluft in hypoxemic patients resuming spontaneous breathing: proportional modes versus pressure support ventilation. Ann Intensive Care. 2023 Dec 20;13(1):131. doi: 10.1186/s13613-023-01230-w. PMID 38117367
- [Background] Bellani G, Grasselli G, Teggia-Droghi M, Mauri T, Coppadoro A, Brochard L, Pesenti A. Do spontaneous and mechanical breathing have similar effects on average transpulmonary and alveolar pressure? A clinical crossover study. Crit Care. 2016 Apr 28;20(1):142. doi: 10.1186/s13054-016-1290-9. PMID 27160458
- [Background] Cornejo RA, Arellano DH, Ruiz-Rudolph P, Guinez DV, Morais CCA, Gajardo AIJ, Lazo MT, Brito RE, Cerda MA, Gonzalez SJ, Rojas VA, Diaz GA, Lopez LDM, Medel JN, Soto DI, Bruhn AR, Amato MBP, Estuardo NR. Inflammatory biomarkers and pendelluft magnitude in ards patients transitioning from controlled to partial support ventilation. Sci Rep. 2022 Nov 23;12(1):20233. doi: 10.1038/s41598-022-24412-1. PMID 36418386
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Background] Su PL, Zhao Z, Ko YF, Chen CW, Cheng KS. Spontaneous Breathing and Pendelluft in Patients with Acute Lung Injury: A Narrative Review. J Clin Med. 2022 Dec 15;11(24):7449. doi: 10.3390/jcm11247449. PMID 36556064
- [Background] Coppadoro A, Grassi A, Giovannoni C, Rabboni F, Eronia N, Bronco A, Foti G, Fumagalli R, Bellani G. Occurrence of pendelluft under pressure support ventilation in patients who failed a spontaneous breathing trial: an observational study. Ann Intensive Care. 2020 Apr 7;10(1):39. doi: 10.1186/s13613-020-00654-y. PMID 32266600
- [Background] Sang L, Zhao Z, Yun PJ, Frerichs I, Moller K, Fu F, Liu X, Zhong N, Li Y. Qualitative and quantitative assessment of pendelluft: a simple method based on electrical impedance tomography. Ann Transl Med. 2020 Oct;8(19):1216. doi: 10.21037/atm-20-4182. PMID 33178748
- [Background] Chi Y, Zhao Z, Frerichs I, Long Y, He H. Prevalence and prognosis of respiratory pendelluft phenomenon in mechanically ventilated ICU patients with acute respiratory failure: a retrospective cohort study. Ann Intensive Care. 2022 Mar 5;12(1):22. doi: 10.1186/s13613-022-00995-w. PMID 35246748
- [Background] Bellani G, Grassi A, Sosio S, Gatti S, Kavanagh BP, Pesenti A, Foti G. Driving Pressure Is Associated with Outcome during Assisted Ventilation in Acute Respiratory Distress Syndrome. Anesthesiology. 2019 Sep;131(3):594-604. doi: 10.1097/ALN.0000000000002846. PMID 31335543
- [Background] Bellani G, Grassi A, Sosio S, Foti G. Plateau and driving pressure in the presence of spontaneous breathing. Intensive Care Med. 2019 Jan;45(1):97-98. doi: 10.1007/s00134-018-5311-9. Epub 2018 Jul 13. No abstract available. PMID 30006893
- [Background] Bastia L, Amendolagine L, Pozzi F, Carenini S, Cipolla C, Curto F, Bellani G, Fumagalli R, Chieregato A. Reliability of Respiratory System Compliance Calculation During Assisted Mechanical Ventilation: A Retrospective Study. Crit Care Med. 2023 Oct 1;51(10):e201-e205. doi: 10.1097/CCM.0000000000005964. Epub 2023 Jun 16. PMID 37326475